CLINICAL TRIAL: NCT04836728
Title: A Randomized, Multicenter, Open-label, Phase II Study of Platinum-Containing Chemotherapy and Sintilimab With or Without Autologous Cytokine-induced Killer Cell Immunotherapy in Stage IV Non-Small Cell Lung Cancer Subjects
Brief Title: Phase II Study of Chemotherapy and PD-1 Inhibitor Combination With Autologous CIK Cell Immunotherapy to Treat Lung Cancer
Acronym: CCICC-002b
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20210014
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Non-small Cell Lung Cancer Metastatic; First-line Treatment
MeSH Terms: interventions — sintilimab; Immune Checkpoint Inhibitors; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CIK cells + Sintilimab + Platinum-based doublet chemotherapy (Experimental): Participants receive CIK cells for up to 8 cycles, in combination with sintilimab plus platinum-based chemotherapy (carboplatin and albumin paclitaxel for squamous NSCLC, or carboplatin and pemetrexed for non-squamous NSCLC), intravenously, every 3 weeks, for up to four cycles, followed by maintenance therapy with sintilimab for squamous NSCLC, and sintilimab plus pemetrexed for non-squamous NSCLC until disease progression or unacceptable toxicity or 2 years.
  Interventions: Biological: CIK cells injection; Drug: Sintilimab Injection; Drug: Pemetrexed; Drug: Albumin paclitaxel; Drug: Carboplatin
- Sintilimab + Platinum-based doublet chemotherapy (Active Comparator): Participants receive sintilimab plus platinum-based chemotherapy (carboplatin and albumin paclitaxel for squamous NSCLC, or carboplatin and pemetrexed for non-squamous NSCLC), intravenously, every 3 weeks, for up to four cycles, followed by maintenance therapy with sintilimab for squamous NSCLC, and sintilimab plus pemetrexed for non-squamous NSCLC until disease progression or unacceptable toxicity or 2 years.
  Interventions: Drug: Sintilimab Injection; Drug: Pemetrexed; Drug: Albumin paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: CIK cells injection — CIK cells, more than 1x10^10 (10 billion ), intravenous infusion, d14, Q3W.
  Other Names: Autologous cytokine-induced killer cells
  Arms: CIK cells + Sintilimab + Platinum-based doublet chemotherapy
Drug: Sintilimab Injection — 200 mg, intravenous infusion, d1, every 3 weeks
  Other Names: PD-1 inhibitor
Drug: Pemetrexed — 500 mg/m^2, intravenous infusion, d1, every 3 weeks
  Other Names: Pemetrexed injection
Drug: Albumin paclitaxel — 260 mg/m^2, intravenous infusion, d1, every 3 weeks
  Other Names: Albumin paclitaxel Injection
Drug: Carboplatin — AUC 5, intravenous infusion, d1, every 3 weeks
  Other Names: Carboplatin injection

SUMMARY:
This prospective, multi-center, open-label, phase II, randomized controlled trial (CCICC-002b) is to evaluate the efficacy and safety of autologous cytokine-induced killer cell immunotherapy in combination with PD-1 inhibitor and platinum-containing chemotherapy in the first-line treatment of stage IV non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any trial-related procedures.
2. Age ≥18 and ≤75 years.
3. Histologically or cytologically confirmed stage IV NSCLC (IASLC/UICC 8th edition TNM staging) with no prior systemic therapy for advanced disease.
4. For enrolled adenocarcinoma patients: Absence of EGFR-sensitive mutations and ALK gene fusion alterations confirmed by histological specimens.
5. At least one radiologically measurable lesion per RECIST v1.1. Lesions within prior radiotherapy fields may be considered measurable if progression is confirmed.
6. No prior systemic antitumor therapy for advanced/metastatic disease. Subjects who received:

   * Platinum-based adjuvant/neoadjuvant chemotherapy, or
   * Definitive chemoradiotherapy for limited-stage disease are eligible if disease progression/recurrence occurred ≥6 months after last chemotherapy.
7. Asymptomatic or stable brain metastases after local treatment are permitted if all criteria are met:

   1. Measurable extracranial lesions
   2. No CNS symptoms or symptom stability for ≥2 weeks
   3. No corticosteroids required, OR discontinued corticosteroids ≥7 days before first dose, OR stable corticosteroid dose ≤10 mg/day prednisone equivalent for ≥7 days.
8. Palliative radiotherapy (including brain RT for symptomatic metastases) is allowed if completed ≥1 week before first dose and radiation-related toxicities have recovered to ≤Grade 1 (CTCAE v5.0, excluding alopecia).
9. ECOG performance status 0-1.
10. Life expectancy >3 months.
11. Adequate organ function meeting all laboratory criteria:

    1. Absolute neutrophil count (ANC) ≥1.5×10⁹/L without granulocyte colony-stimulating factor support within 14 days.
    2. Platelets ≥100×10⁹/L without transfusion within 14 days.
    3. Hemoglobin >9 g/dL without transfusion or erythropoietin within 14 days.
    4. Total bilirubin ≤1.5×ULN.
    5. AST/ALT ≤2.5×ULN (≤5×ULN if liver metastases present).
    6. Serum creatinine ≤1.5×ULN AND creatinine clearance (Cockcroft-Gault formula) ≥60 mL/min.
    7. INR/PT ≤1.5×ULN.
    8. Normal thyroid function (TSH within normal range). Subjects with baseline TSH outside normal range may enroll if FT3/FT4 are normal.
    9. Normal myocardial enzyme profile.
12. For women of childbearing potential: Negative urine/serum pregnancy test within 3 days prior to first dose (Cycle 1 Day 1). Non-childbearing potential is defined as ≥1 year post-menopause, surgically sterilized, or hysterectomy.
13. All subjects (regardless of gender) at risk of conception must use highly effective contraception (failure rate <1% annually) during treatment and for 120 days (or 180 days per protocol) after last dose.

Exclusion Criteria:

1. Pathologically confirmed small cell lung cancer (SCLC), including mixed SCLC-NSCLC histology.
2. Prior radiotherapy meeting any of the following:

   1. Radiation to ≥30% of bone marrow within 14 days before first dose
   2. Lung radiation >30 Gy within 6 weeks before treatment (subjects must have recovered to ≤Grade 1 toxicity, no corticosteroid requirement, and no history of radiation pneumonitis)
   3. Palliative radiotherapy completed ≤7 days before first dose
3. Diagnosis of malignancies other than NSCLC within 5 years before first dose (except cured basal cell carcinoma, squamous cell carcinoma, or resected carcinoma in situ).
4. Current participation in interventional clinical trials or receipt of investigational drugs/devices within 4 weeks before first dose.
5. Prior therapy with anti-PD-1/PD-L1/PD-L2 agents or drugs targeting other T-cell co-stimulatory/checkpoint pathways (e.g., CTLA-4, OX-40, CD137).
6. Systemic treatment with Chinese herbal medicines (for lung cancer indications) or immunomodulatory agents (e.g., thymosin, interferon, interleukin) within 14 days before first dose (except local pleural control).
7. Active autoimmune disease requiring systemic treatment (e.g., disease-modifying agents, corticosteroids, immunosuppressants) within 2 years before first dose. Replacement therapies (e.g., thyroid hormone, insulin, physiologic corticosteroids) are permitted.
8. Systemic corticosteroids (>10 mg/day prednisone equivalent) or immunosuppressive therapy within 7 days before first dose (excluding topical/nasal/inhaled corticosteroids).

   *Note: Physiologic corticosteroid doses (≤10 mg/day prednisone equivalent) are allowed.*
9. Clinically uncontrolled pleural/peritoneal effusion (subjects with stable effusion not requiring drainage or ≥3 days post-drainage may enroll).
10. History of allogeneic organ transplantation (except corneal transplants) or hematopoietic stem cell transplantation.
11. Known hypersensitivity to sintilimab, pemetrexed, nab-paclitaxel, carboplatin, or their excipients.
12. Failure to recover from prior intervention-related toxicities (≤Grade 1 or baseline, excluding alopecia/fatigue) before treatment initiation.
13. Known HIV infection (HIV 1/2 antibody positive).
14. Untreated active hepatitis B (HBsAg-positive with HBV-DNA > upper limit of normal [ULN] at local laboratory).

    *Exceptions:*
    1. HBV-DNA <1000 copies/ml (200 IU/ml) before first dose with ongoing antiviral prophylaxis during chemotherapy
    2. Anti-HBc(+) subjects with HBsAg(-), anti-HBs(-), and undetectable HBV-DNA may enroll without prophylaxis but require close monitoring
15. Active HCV infection (HCV antibody-positive with detectable HCV-RNA).
16. Live vaccination within 30 days before Cycle 1 Day 1. *Note: Inactivated vaccines (e.g., seasonal influenza) are permitted; live attenuated vaccines (e.g., nasal flu vaccine) are prohibited.*
17. Pregnancy or lactation.
18. Severe uncontrolled systemic diseases including:

    1. Symptomatic ECG abnormalities (e.g., complete left bundle branch block, ≥Grade 2 AV block, ventricular arrhythmias, atrial fibrillation)
    2. Unstable angina, congestive heart failure (NYHA class ≥2)
    3. Myocardial infarction within 6 months
    4. Poorly controlled hypertension (SBP >140 mmHg/DBP >90 mmHg)
    5. Non-infectious pneumonitis requiring steroids within 1 year or active interstitial lung disease
    6. Active tuberculosis
    7. Uncontrolled active infection requiring systemic therapy
    8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction
    9. Decompensated liver disease (e.g., cirrhosis, active hepatitis)
    10. Poorly controlled diabetes (fasting glucose >10 mmol/L)
    11. Urine protein ≥++ with 24-hour protein >1.0 g
    12. Uncontrolled hypercalcemia (>1.5 mmol/L ionized calcium or corrected serum calcium >ULN)
    13. Non-healing wounds/fractures
    14. Psychiatric disorders impairing protocol compliance
19. Any condition that may interfere with study results, compromise subject safety, or preclude full participation as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Time Frame: Up to 24 months
  ORR was defined as the percentage of patients with a confirmed complete (CR) or partial response (PR) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the investigator.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  PFS was defined as the time from the initial treatment to the first occurrence of disease progression or all-cause death (whichever occurs first) assessed by the investigator according to RECIST v1.1.
Overall Survival (OS) | up to 3 years
  OS was defined as the time from the initial treatment until the date of death due to any cause.
Duration of response (DOR) | up to 24 months
  DOR was defined as first documented evidence of a CR or PR until PD or death as determined by the investigator according to RECIST v1.1.
Disease Control Rate (DCR) | up to 24 months
  DCR was defined as the proportion of patients with the best overall response of CR, PR, and stable disease (SD) as determined by the investigator according to RECIST 1.1.
Number of Participants Who Experienced an Adverse Event (AE) | up to 24 months (Serious AEs: Up to 90 days after last dose of study treatment (Other AEs: Up to 30 days after last dose of study treatment)
  An AE was defined as any untoward medical occurrence in a study participant administered with study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who experienced an AE is presented.
Number of Participants Who Discontinued Any Study Drug Due to an AE | up to 24 months
  An AE was defined as any untoward medical occurrence in a study participant administered with study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who discontinued any randomized study drug due to an AE is presented.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Liu, MD. Ph.D, Study Director — Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
This is a multicenter, prospective clinical trial. Eight centers provide data to each other.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: All patients